CLINICAL TRIAL: NCT04119349
Title: Influence of Prenatal Counseling on the Attitudes and Preferences Towards Invasive Prenatal Testing Among Women in Their First Trimester of Pregnancy
Brief Title: Influence of Prenatal Counseling in Invasive Testing
Acronym: INVASIVE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital Clinic of Barcelona (Other)
Responsible Party: Principal Investigator, Raigam Jafet Martinez Portilla, Principal investigator, Hospital Clinic of Barcelona
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: IRN2019/03/0001
Record Dates: First submitted 2019-10-04; First posted 2019-10-08 (Actual); Last update posted 2019-11-13 (Actual); Status verified 2019-11

CONDITIONS: Genetic Counseling; Prenatal Diagnosis

STUDY DESIGN:
Intervention Model Description: Participants will be randomized using an interactive Web-response system assigning patients in a 1:1 ratio to receive the extra counseling before first trimester assessment (intervention group) or nothing (control group). The allocation will be performed by the study manager. The maternal-fetal medicine specialist will be in charge of the participant's enrolment and will also perform the intervention to the corresponding randomized group.
  This is an open-label study which means that the specialist and women will be aware of the allocation and intervention every time.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Counseling (Experimental): Women are given extra 15-minute counseling on the pros and cons of all different methods for prenatal testing including no testing at all
  Interventions: Behavioral: Extra counseling
- Standard care (No Intervention): Women receiving standard care by means of counseling

INTERVENTIONS:
Behavioral: Extra counseling — Participants will be given an extra 15-minute prenatal counseling before their first-trimester scan. The extra counseling, which is the intervention in the experimental group, consists of an explanation of all screening techniques for chromosomal abnormalities, including the first trimester combined test, cfDNA testing, invasive testing, and no screening at all.
  Arms: Counseling

SUMMARY:
It is well established that screening for Down syndrome should be offered in the first trimester to each pregnant woman. The most common screening method is nowadays the first trimester combined test which consists of a Bayesian analysis of the a priori risk of maternal age for Down's syndrome, and the posterior risk combining serum biomarkers such as beta fraction of the human chorionic gonadotropin (β-hCG), pregnancy-associated plasma protein-A (PAPP-A), and nuchal translucency measurement. Women at high risk for trisomy 21 or 18 using this combined test are eligible for chorionic villous sampling or amniocentesis for a final diagnosis. In recent years there has been a huge advance in prenatal screening for Down's syndrome with the advent of cell free DNA testing with higher sensitivity and specificity than the combined test, in which a positive result must be also confirmed by an invasive diagnostic procedure. But as the range of options broadens, also the need for health education to allow women to have an adequately informed decision process on which prenatal test better suits their needs. In multicultural cities, this has become especially important to integrate patient's values and expectations to an evidence-based decision regarding prenatal testing. There is high-quality evidence demonstrating that aversion to risk of fetal loss related to an invasive test may come from incomplete information, shaping the attitude towards which test to choose from the mother's point of view. And the disbelief that by taking cfDNA testing the risk of miscarriage would be reduced.

Many information is available about preferences and attitudes in prenatal testing from Northern European studies, but scarce information is available from Southern Europe, where the amniocentesis rate in the nineties was as high as 40% of the urban pregnant population.

The investigators hypothesize that when enough information is given before the initial screening, women will overcome aversion to invasive testing and will be more likely to choose this method as their first choice when compared to women having routine care.

DETAILED DESCRIPTION:
Study design:

This is a randomized open-label controlled trial evaluating the impact of an extra 15-minute prenatal counseling before the first trimester combined screening test for Down's syndrome, on the women's attitudes and preferences towards having invasive testing as the first-line option for the screening of chromosomal abnormalities.

Data will be collected by the study-site manager and stored in an electronic data-capture database. The coordinator of the study and the statistician will witness the accuracy of the data at the beginning, middle, and end of the study (on-site audit). Data will be captured in a paper form basis and then captured into the electronic database.

Sample size calculation has been made using an independent two-sample proportions likelihood-ratio test. The investigators expect a 10% of women willing to have an invasive procedure as a first-line test for aneuploidies in the control group, and a 25% difference to those in the experimental group that is given an extra 15-minute prenatal counseling, this yields a sample of 42 women per arm with a total of 84 subjects using a Type I error of 0.0501 and a power of 80% by a two-sided test.

Randomization and intervention

Questionnaire The questionnaire consists of twenty-one questions assessing the knowledge, preferences, and attitude towards prenatal testing in the first trimester of pregnancy. The questionnaire will be divided into two parts. The first fourteen questions consist of demographic characteristics and obstetrics history, such as age, ethnicity, study level, marital status, religion, salary, employment, parity, previous miscarriages, previous terminations of pregnancy, previous congenital defects, pregnancy search time in months, type of conception, and who had provided any type of previous information about prenatal screening/testing. Women will be asked to select only one option for each question. All questions will have the possibility to answer as "Prefer not to answer". The second part of the questionnaire will assess the preferences and attitudes towards prenatal testing; women will be asked to choose only one option for each question. The following questions will be included in the second part of the questionnaire: What influences the participants the most about prenatal testing? Who influenced the participants the most about prenatal testing? Would the participants like to choose their prenatal test? Which prenatal test would the participants choose? What is the participants' opinion about termination? All questions include an "I don't know answer". The two final questions will ask the following, "What information regarding the results of prenatal testing is more important for the participants?" and "What is most important for the participants about prenatal testing?". Women will be asked to score the first question from 1 to 5, meaning 1 the least important and 5 the most important, and from 1 to 6 in the same manner for the second question. These two questions will be assessed as means, where the question with the highest mean represents what is most important for the patient.

The analysis will be conducted by intention-to-treat. Missing data for the main outcome will be handled by complete-data analysis because women without an answer on the main outcome will be excluded. All analyses will be divided by groups (control vs experimental group). Continuous data will be assessed for normality using the Kolmogorov-Smirnoff test. Normally distributed variables will be compared using t-test and expressed as mean and standard deviation (SD), while not normally distributed variables will be analyzed using the Mann-Whitney-U test and expressed as medians and interquartile range (IQR). Quantitative variables will be compared using X2 test and expressed as numbers (n) and proportions (%). For the main outcome, preferences for prenatal testing among groups will be analyzed using absolute risk increase defined as the incidence of the outcome in the experimental group minus the incidence in the control group. The absolute risk increase will be depicted in a forest plot. A multivariate logistic regression will be performed to determine the Odds for choosing invasive testing adjusting by demographic characteristics and previous counseling. Data will be analyzed using STATA v.15.3 for Mac (Texas College Station) and GraphPad Prism version 8.1.2 for Mac, GraphPad Software, San Diego, California USA, www.graphpad.com.

ELIGIBILITY:
Inclusion Criteria:

* any pregnant woman attending the first trimester combined screening test for chromosomal abnormalities
* Singleton or twin pregnancies
* Between 11+0 and 13+6 weeks' gestation

Exclusion Criteria:

* women not willing to participate in the study
* women without an answer in the question regarding which prenatal test would they choose (main outcome)
* women with no sufficient knowledge of Spanish or Catalan to be able to read and understand the questionnaire

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2019-10-10 (Actual); Primary Completion 2019-11-11 (Actual); Study Completion 2019-11-11 (Actual)

PRIMARY OUTCOMES:
Preference for an invasive testing | Through study completion, an average of 1 month
  The primary outcome of the study is the desire to choose an invasive diagnostic testing as the first option of screening for chromosomal abnormalities.
  This will be measured in the questionnaire by asking the question: which prenatal test would you choose if given the opportunity? Women will be asked to choose only one answer between first trimester combined test, cell-free DNA, invasive testing in a yes/no format. The main outcome will be analized as the absolute risk increase along with tis 95% confidence interval.

CONTACTS AND LOCATIONS:
Overall Officials: Raigam J MartinezcPortilla, MD, Principal Investigator — Hospital Clinic of Barcelona
Locations (1):
- Hospital Clinic of Barcelona, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Paz Y Mino F, Martinez-Portilla RJ, Pauta M, Borrell A. A Randomized Controlled Trial on the Influence of Prenatal Counseling on the Attitudes and Preferences Toward Invasive Prenatal Testing Among Women in Their First Trimester of Pregnancy (INVASIVE). Front Genet. 2020 Nov 9;11:561283. doi: 10.3389/fgene.2020.561283. eCollection 2020. PMID 33240315

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-09-15): https://cdn.clinicaltrials.gov/large-docs/49/NCT04119349/Prot_SAP_000.pdf